CLINICAL TRIAL: NCT01428752
Title: Prevalence of Colorectal Adenoma in 30- to 49-year-old Asymptomatic Subjects With a First Relative History of Colorectal Cancer
Brief Title: Study of Prevalence of Colorectal Adenoma in 30- to 49-year-old Subjects With a Family History of Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jaeil Kim, Clinical Assistant Professor, Asan Medical Center
Other Study IDs: ADENOMA 30-49 YO
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Colorectal Neoplasms
Keywords: colonoscopy; colorectal neoplasms; screening; family history
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood and serum Colorectal polyp/cancer tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Family history: 30- to 49-year-old asymptomatic subjects with a first relative history of colorectal cancer

SUMMARY:
Current guidelines for initiating screening colonoscopies in patients younger than 50 years of age who have a first relative history of colorectal cancer are controversial. The aim of this study was to prospectively define the prevalence of colorectal adenoma 30- to 49-years-old asymptomatic subjects with a first relative history of colorectal cancer and to compare the data with controls.

Design: Single-center prospective study

DETAILED DESCRIPTION:
Colorectal cancer screening is recommended for average-risk persons beginning at age 50. A family history of colorectal cancer is recognized as a risk factor for colorectal adenoma. However, the strength of this association is uncertain. Current guidelines for initiating screening colonoscopies in patients younger than 50 years of age who have a first relative history of colorectal cancer have proved controversial. The conflicting recommendations are partly attributable to the lack of data about the prevalence of CRC and adenomas among 30- to 49-year-old individuals with a first relative history of colorectal cancer. This prospective study will quantify the prevalence of adenomas (any size) and advanced adenomas among 30- to 49-year-old individuals undergoing their first screening colonoscopy because of a first relative history of colorectal cancer and compare the data with controls(asymptomatic subjects without a first relative history of colorectal cancer).

ELIGIBILITY:
Inclusion Criteria:

* 30- to 49-year-old asymptomatic subjects
* First relative history of colorectal cancer

Exclusion Criteria:

* previous colonoscopy for any reason
* personal history of colorectal adenomas or CRC
* history of familial adenomatous polyposis, hereditary nonpolyposis colorectal cancer, or inflammatory bowel disease
* documented history of occult GI bleeding, lower gastrointestinal tract bleeding not attributable to hemorrhoid, or
* iron deficiency anemia
* unexplained weight loss of >10% of the body weight in the 6 months before colonoscopy
* incomplete examination of entire colon

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 30- to 49-year-old asymptomatic subjects undergoing first screening colonoscopy because of a first relative history of colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
prevalence of colorectal adenoma(any size) | First screening colonoscopy

SECONDARY OUTCOMES:
prevalence of advanced adenoma | First screening colonoscopy
  1. Any adenoma ≥10 mm
  2. Any villous component
  3. High-grade dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Jo Kim, M.D, Study Director — Department of Gastroenterology, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea